CLINICAL TRIAL: NCT01631422
Title: Single-Center, Open-label Study Investigating the Excretion Balance, Pharmacokinetics and Metabolism of a Single Oral Dose of [14C]-Radio-labeled RO4602522 in Healthy Male Volunteers
Brief Title: A Single Dose Study of Radiolabeled RO4602522 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: BP28235; 2012-000587-26 (EudraCT Number)
Record Dates: First submitted 2012-06-20; First posted 2012-06-29 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — sembragiline

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: RO4602522

INTERVENTIONS:
Drug: RO4602522 — Single radiolabeled dose

SUMMARY:
This single-center, open-label study will investigate the pharmacokinetics and elimination of a radiolabelled dose of RO4602522 in healthy male volunteers. The healthy male volunteers will receive a single oral dose of RO4602522.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, 35 to 55 years of age, inclusive
* Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead electrocardiogram (ECG), hematology, blood chemistry, serology and urinalysis
* A body mass index (BMI) between 18 to 30 kg/m2 inclusive
* Male volunteers and their partners of childbearing potential must use 2 methods of contraception, one of which must be a barrier method for the duration of the study and for 90 days after the last dose.
* Able to participate and willing to give written informed consent and to comply with the study restrictions.
* Non-smokers or have not smoked since at least 3 months prior to screening

Exclusion Criteria:

* If capable of reproduction, unwilling to use an effective form of contraception
* Suspicion of regular consumption of drug of abuse and/or positive drug or alcohol screen
* Infection with hepatitis B, hepatitis C, or human immunodeficiency virus 1 and 2
* Systolic blood pressure greater than 140 or less than 90 mm Hg, and diastolic blood pressure greater than 90 or less than 50 mm Hg
* Resting pulse rate greater than 90 or less than 45 beats per minute
* Clinically significant abnormalities in laboratory test results
* Participation in an investigational drug or device study within 90 days prior to screening
* Donation of blood within 3 months prior to screening
* Concomitant disease or condition that could interfere with, or treatment of which might interfere with, the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2012-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Elimination of RO4602522: urine/feces concentration | Predose, Day 1, 2 and 3
Pharmacokinetics: Plasma concentration of RO4602522/metabolite | Predose, Day 1, 2 and 3

SECONDARY OUTCOMES:
Pharmacokinetics: Metabolic profile of RO4602522: plasma/urine/feces concentration | Predose, Day 1, 2 and 3

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Zuidlaren, Netherlands